CLINICAL TRIAL: NCT06498388
Title: Building the Predictive Model of the BRA-based ViscoElastography (BRAVE) System for Detecting Breast Cancer Tumors (BRAVE Discovery Study)
Brief Title: Predicting Breast Cancer With the BRAVE System
Acronym: BRAVE
Status: Recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Cancer Research Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-5453
Record Dates: First submitted 2024-06-03; First posted 2024-07-12 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Breast Mass; Breast Cancer
Keywords: Breast mass; Breast cancer; Mammogram; Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal Mammographic Breast Density (NMBD): Women with Normal Mammographic Breast Density (NMBD): Each participant will take part in one imaging session, using the BRAVE system.
  Interventions: Other: Stiffness measurement by visco-elastography
- Elevated Mammographic Breast Density (EMBD): Women with Elevated Mammographic Breast Density (EMBD): Each participant will take part in one imaging session, using the BRAVE system.
  Interventions: Other: Stiffness measurement by visco-elastography

INTERVENTIONS:
Other: Stiffness measurement by visco-elastography — Participant will be asked to put on the study's bra with the help of a female member of the team if necessary and to complete the examination process.

SUMMARY:
Breast cancer predominates among cancer diagnoses in Canadian women. It accounts for around 25% of new cases and contributes to 13% of all cancer-related deaths. In 2020, almost 27,400 Canadian women were diagnosed with breast cancer and 5,000 of them died from it.

Mammography is still the preferred method for screening for breast cancer. Although progress has been made over the years, mammography does have its drawbacks. These include physical discomfort for patients, exposure to X-rays and reduced effectiveness in dense breasts. The study team is therefore interested in developing a new breast cancer detection method, the BRAVE method.

The BRAVE method, short for "BRA-based Visco-Elastography", uses the high contrast of elastic stiffness in malignant breast tumors to detect possible cancer cases without the need for X-rays or breast compression.

The first phase, carried out on a small scale pilot study, aimed to assess the method's ability to distinguish a breast with no abnormalities from one with confirmed cancer. The second phase (current phase), carried out on a larger scale, aims to confirm the sensitivity and specificity of the method in detecting malignant lesions, i.e. to determine whether the method is capable of distinguishing between several types of breast masses.

DETAILED DESCRIPTION:
This study has two objectives, which will be studied in two separate groups.

1. To measure the sensitivity and specificity of BRAVE in identifying malignant lesions in a cohort of 300 women.
2. To assess the impact of breast density on the ability of BRAVE to discriminate malignant breast lesions.

The research team aim to recruit 300 women requiring follow-up imaging. Half will have lower breast density (categories A or B) and the other half will have higher breast density (categories C or D).

Participants will need to attend a single visit lasting approximately 75 minutes, where they will be asked to wear the study's bra and complete the examination process.

Other data will also be collected in the medical file to enable the team to confirm: the density of the breast, and the results and dates of mammography imaging or other tests related to breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Able and willing to provide signed informed consent in French or English
* Recent mammogram (< 6 months)
* Breast mass newly identified by palpation, mammography, sonography, or MRI and have been referred for additional imaging or evaluation.

Specific inclusion Criteria:

Group 1 - Normal Mammographic Breast Density (NMBD): Breast density A or B Group 2 - Elevated Mammographic Breast Density (EMBD): Breast density C or D

Exclusion Criteria:

* Pregnant or breast-feeding women
* Breast implants or prior surgery/biopsy to breasts
* Any disease or condition limiting the capacity to complete the examination process
* Any previous or prescribed treatment against cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 ≥18 years old women with a recent mammogram and a reference for additional imaging or evaluation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Stiffness of the breasts | Once, at recruitment, up to 6 months after mammography
  Main marker that will be assessed for its capacity to identify malignant lesions. It will be measured by the viscoelastic property values determined by the BRAVE system.
Risk and malignancies lesions (RnMLs) | At the time of mammogram, which will be no more than 6 months prior to recruitment
  Defined by mammography, additional imaging and biopsy results and scored as BI-RADS 5 to 6.

SECONDARY OUTCOMES:
Breast density | Once, at mammogram (up to 6 months prior to recruitement)
  The breast density can be scored as A: low-density, B: few areas of dense tissue, C: evenly dense, D: extremely dense, and is determined by standard of care imaging. Participants will be gathered in either NMBD group (A or B; normal density) or EMBD group (C or D, elevated density).

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Van Houten, PhD, ing., Principal Investigator — Université de Sherbrooke
Locations (1):
- CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No